CLINICAL TRIAL: NCT06283563
Title: The Effect of Online Physical Activity Tracking on Physical Activity Level, Psychological Health, Fatigue and Quality of Life in Patients With Multiple Sclerosis
Brief Title: Online Physical Activity Tracking in Patients With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/5474
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: physical activity; depression; life quality; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive reminders regarding physical activity promotion via the social media group created.
  Interventions: Other: Physical activity tracking
- Control group (Active Comparator): Participants will be encouraged to continue their routine lives.
  Interventions: Other: No physical activity tracking

INTERVENTIONS:
Other: Physical activity tracking — At the beginning, patients will be given a brief information about the benefits of exercise training. Additionally, a short brochure explaining the effects of exercise in MS will be given. Participants in the intervention group will be asked to join one of two groups created by the researchers via messaging app. Reminders will be arranged on Monday-Wednesday-Thursday in one of the groups, and on Tuesday-Thursday-Saturday in the other group. In this regard, it will be emphasized that he/she should exercise at least 3 days a week. In this regard, they will be encouraged to walk for at least 30 minutes, 3 days a week, on the days they determine. The total intervention period will be 8 weeks. Reminders to exercise will be given by the researchers in the created messaging app group. Patients will be reminded to take their mobile phones with them during physical activity and to record their daily exercise minutes.
  Arms: Experimental group
Other: No physical activity tracking — At the beginning, patients will be given a brief information about the benefits of exercise training. Additionally, a short brochure explaining the effects of exercise in multiple sclerosis will be given. Participants will be encouraged to continue their routine lives and no reminders will be given.
  Arms: Control group

SUMMARY:
This study aims to investigate the effects of regular remote monitoring of physical activity levels of individuals with multiple sclerosis on physical activity levels, psychological health, fatigue and quality of life.

DETAILED DESCRIPTION:
The study population will consist of patients with multiple sclerosis. Participants in the intervention and control groups will initially be given a brief briefing about the benefits of exercise training. Additionally, a short brochure explaining the effects of exercise in multiple sclerosis will be given. Participants in the intervention group will be allowed to join the group created by the researchers via Whatsapp. In this regard, it will be emphasized that should exercise at least 3 days a week. The participant will be asked to fill out the survey created via Google form in order to record their activity minutes in these three days. The total intervention period will be 8 weeks. Reminders to exercise will be given by the researchers in the created Whatsapp group. Participants in the control group will be encouraged to continue their routine lives. Average step counts will be recorded before and after treatment. Additionally, they will be asked to report their average step count each week via WhatsApp groups. Pre- and post-intervention evaluations will be carried out by a physiotherapist. Patients' physical activity levels, depression and anxiety, fatigue and quality of life parameters will be examined.

ELIGIBILITY:
Inclusion Criteria:

->18 years old

* Being diagnosed with multiple sclerosis according to McDonald's diagnostic criteria, owning a smartphone and using the WhatsApp application,
* Having regular internet access
* Not participating in a regular physical activity program in the last 6 months,
* Expanded Disability Status Scale<6

Exclusion Criteria:

* Having an attack during work,
* Any orthopedic or neurological disorder that affects compliance with the physical activity program,
* Not having independent mobility ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Smartphone pedometer | Baseline
  The number of steps in the pedometer application of the current smartphone on the individual's phone will be recorded.
Smartphone pedometer | 8 week
  The number of steps in the pedometer application of the current smartphone on the individual's phone will be recorded.
International Physical Activity Questionnaire - Short Form | Baseline
  It consists of 8 questions with a recall period defined as 'last week'. The questions of the scale ask whether the participant walks for at least 10 minutes on any given day or does moderate or vigorous activities, and how much time/day the individual spends on each of these activities.
International Physical Activity Questionnaire - Short Form | 8 week
  It consists of 8 questions with a recall period defined as 'last week'. The questions of the scale ask whether the participant walks for at least 10 minutes on any given day or does moderate or vigorous activities, and how much time/day the individual spends on each of these activities.

SECONDARY OUTCOMES:
Beck Depression Inventory II | Baseline
  Inventory consists of 21 items, in which four response options are presented on a scale of 0 to 3. For example, to measure pessimism (item 2) the response options used range from "I am not particularly discouraged about the future" (score of 0) to "the future is hopeless and things cannot improve" (score of 3).
Beck Depression Inventory II | 8 week
  Inventory consists of 21 items, in which four response options are presented on a scale of 0 to 3. For example, to measure pessimism (item 2) the response options used range from "I am not particularly discouraged about the future" (score of 0) to "the future is hopeless and things cannot improve" (score of 3).
Beck Anxiety Inventory | Baseline
  The Beck Anxiety Inventory consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Beck Anxiety Inventory | 8 week
  The Beck Anxiety Inventory consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Fatigue Severity Scale | Baseline
  The classification is <36 mild no fatigue, 36-52 = moderate fatigue and >52 severe fatigue
Fatigue Severity Scale | 8 week
  The classification is <36 mild no fatigue, 36-52 = moderate fatigue and >52 severe fatigue
Multiple Sclerosis Quality of Life-54 | Baseline
  It is a multidimensional, health-related quality of life measure that combines both general and MS-specific items into a single instrument. It consists of a total of 54 items. Patients will be considered to have a better quality of life as they get closer to 100 on a 0-100 rating system.
Multiple Sclerosis Quality of Life-54 | 8 week
  It is a multidimensional, health-related quality of life measure that combines both general and MS-specific items into a single instrument. It consists of a total of 54 items. Patients will be considered to have a better quality of life as they get closer to 100 on a 0-100 rating system.

CONTACTS AND LOCATIONS:
Overall Officials: BURCU talu, Study Director — Inonu University

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared with other researchers if desired.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study was published
Access Criteria: If requested from the authors, it can be shared with researchers at the authors' discretion.